CLINICAL TRIAL: NCT01311830
Title: Enhancing Smoker Utilization of the Minnesota Quitline Through Support Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: ClearWay Minnesota (Unknown)
Responsible Party: Christi Patten, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-005379
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Counseling (Active Comparator)
  Interventions: Behavioral: Telephone Counseling
- Written Materials (Placebo Comparator)
  Interventions: Behavioral: Written Materials

INTERVENTIONS:
Behavioral: Telephone Counseling
  Arms: Telephone Counseling
Behavioral: Written Materials
  Arms: Written Materials

SUMMARY:
This study will develop an intervention for adults who want to support a smoker. The goal of the intervention is for the support person to motivate & encourage their smoker to call the state Quitline funded by Minnesota ClearWay. The study will examine the efficacy of a telephone based intervention for support persons compared to a self-help intervention (written materials only).

DETAILED DESCRIPTION:
To have the greatest impact on the public health, interventions need to reach as large a proportion of the smoking population as possible. A significant science base now exists that demonstrates the effectiveness of tobacco quitlines. While the provision of telephone counseling has improved the reach of treatment services to smokers, research is needed to enhance their utilization or reach. In 2001, ClearWay Minnesota (formerly known as MPAAT [Minnesota Partnership for Action Against Tobacco) funded the QUITPLAN Helpline, a telephone-based tobacco cessation counseling service for Minnesotans. Consistent with findings from other quitlines, the QUITPLAN Helpline has reached only 1.5% of smokers in Minnesota. Nonsmokers have a substantial potential role in tobacco control efforts. They represent 82% of the adult population of Minnesota. A novel approach to increasing smoker utilization of effective cessation services is by focusing on nonsmokers who want to help a smoker, i.e., support persons or proxies. Numerous studies provide evidence for the role of extra-treatment social support in smoking cessation. The current study builds on our previous work which indicated the feasibility and potential efficacy of directly recruiting and providing intervention for support persons. Cohen?s theory of social support and health is the conceptual basis for the proposed intervention.

In the first phase of this study, we will pilot the intervention to obtain support person feedback in refining the telephone counseling and other study procedures. We will recruit 30 nonsmoking adult support persons for the pilot to complete the 3-session telephone counseling intervention. Assessments will be completed by mail at baseline and week 4. In phase 2, after refining the intervention, we will use a randomized, two-group design to examine the effect of a 3-session telephone-based intervention versus a self-help intervention (written materials) for nonsmoking adult support persons on increasing their smokers? utilization of the ClearWay Minnesota funded QUITPLAN Helpline. Repeated mailed assessments will be completed by support persons at baseline (week 0) and follow-up at weeks 4 and 26. This study, funded by ClearWay Minnesota, addresses their funding priority area to ?Increase the Availability and Use of Individual Cessation Services.? The Primary Aims of phase 2 are (1) To determine if providing the telephone-based intervention for nonsmoking adult support persons results in a greater proportion of their smokers who call the QUITPLAN Helpline compared to the self-help intervention over the 26 week study period; and (2) To compare treatment groups on change in supportive behaviors provided (Support Provided Measure score) from baseline to week 4. Secondary Aims are to compare the smoker's readiness to quit and utilization of cessation service in the two groups.

We will recruit 564 (30 phase 1, 534 phase 2) nonsmoking adult support persons throughout the entire state of Minnesota using mass media and outreach approaches. They must be interested in supporting a current cigarette smoker who is 18 years of age or older and a resident of Minnesota. In phase 2, support persons will be randomly assigned to receive written self-help materials only (N=237; control group) or to receive the same written materials plus three, 15-20minute telephone-based sessions (N=237; experimental group) stratified according to whether or not the support person lives in the same residence as their smoker. The written materials will be mailed to the support person?s home. These materials will include a QUITPLAN Helpline toll-free number developed specifically for this study and a study reference code that reflects the support person's group assignment and includes the support person?s study ID number (e.g., BLUE 012) that the smoker should provide to the QUITPLAN Helpline intake staff if and when he/she decides to call. The primary dependent variable will be the proportion of support persons? smokers who call the QUITPLAN Helpline anytime during the interval from randomization through week 26, documented by the QUITPLAN Helpline intake staff. (using the study reference code).

The chi-square test will be used to examine treatment differences on the proportion of support persons whose smokers called the QUITPLAN Helpline at least once between randomization into the study and week 26 (Primary Aim 1). Additionally, the two groups will be compared on the time of the smoker?s first call using the Kaplan-Meier method with a log rank test. Support persons whose smoker does not call the Helpline will be censored at week 26. The mean change in Support Provided Measure total score at weeks 4 and 26 will be compared between treatment groups using a two-sample t-test (Primary Aim 2). For each dependent variable, a secondary analysis, using logistic regression or analysis of covariance as appropriate, will be performed to assess treatment effects adjusting for any baseline characteristics that are found to differ between groups.

ELIGIBILITY:
Inclusion Criteria:

1. reside in Minnesota
2. be 18 years of age or older
3. provide written informed consent
4. be a never or former cigarette smoker (no cigarette smoking in the past 6 months)
5. be interested in supporting a current cigarette smoker (has smoked a total of >1 cigarettes during the past 7 days) who is 18 years of age or older and who resides in Minnesota
6. be able and willing to participate in all aspects of the study
7. have access to a working telephone
8. have current and anticipated contact (any combination of face-to-face, telephone, or electronic mail) with the smoker on at least 3 days a week for the 26 week study duration.

Individuals will be excluded if another support person from the same household has enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
proportion of smokers in each group who call the Minnesota Quitline, and changes in supportive behaviors among the support persons as measured by the Support Provided Measure. | 6 months

SECONDARY OUTCOMES:
quit attempts and changes in readiness to quit among the smokers | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Patten CA, Smith CM, Brockman TA, Decker PA, Hughes CA, Nadeau AM, Sinicrope PS, Offord KP, Lichtenstein E, Zhu SH. Support-person promotion of a smoking quitline: a randomized controlled trial. Am J Prev Med. 2011 Jul;41(1):17-23. doi: 10.1016/j.amepre.2011.03.012. PMID 21665059